CLINICAL TRIAL: NCT02731430
Title: Intrathecal Morphine for Postoperative Pain Management in Patients Undergoing Laparoscopic Bariatric Surgery
Brief Title: Intrathecal Morphine for Postoperative Analgesia Following Laparoscopic Bariatric Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Mohammad Abd El-Rahman, Lecturer of anesthesia, icu, and pain management, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 274
Record Dates: First submitted 2016-04-03; First posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group I: morphine group (Active Comparator): received 0.3mg morphine (0.3ml) added to 1.2ml of bupivacaine 0.5% (total volume 1.5ml), intrathecally, immediately before induction of general anesthesia.
  Interventions: Drug: intrathecal morphine
- group II: control group (Placebo Comparator): received 0.3ml saline added to 1.2mlof bupivacaine 0.5% (total volume 1.5ml), intrathecally, immediately before induction of general anesthesia.
  Interventions: Drug: intrathecal saline

INTERVENTIONS:
Drug: intrathecal morphine — received 0.3mg morphine (0.3ml) added to 1.2ml of bupivacaine 0.5% (total volume 1.5ml), intrathecally, immediately before induction of general anesthesia.
  Arms: group I: morphine group
Drug: intrathecal saline — received 0.3ml saline added to 1.2mlof bupivacaine 0.5% (total volume 1.5ml), intrathecally, immediately before induction of general anesthesia.
  Arms: group II: control group

SUMMARY:
this study compares the use of intrathecal morphine, to multimodal analgesic techniques for postoperative pain management following laparoscopic bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia (ASA) II-III patients.
* Aged 30-50 years.
* The body mass index (BMI) of the patients needed to be over 40 kg/m² or over 35 kg/m² with at least one comorbidity.

Exclusion Criteria:

* Patients with a known allergy to the study drugs.
* Advanced cardiac, respiratory, renal or hepatic disease.
* Coagulation disorders.
* Infection at or near the site of intrathecal injection.
* Drug or alcohol abuse.
* Psychiatric illnesses that may interfere with perception and assessment of pain.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Total postoperative analgesic consumption. | 24 hours postoperative
  the efficacy of the studied dose of intrathecal morphine in reducing postoperative analgesic consumption.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) scores | 24 hours postoperative
  postoperative pain scores
Time to first request of rescue analgesia. | 24 hours postoperative
Tolerability as assessed by the incidence of side effects | 24 hours postoperative
  the incidence of side effects

IPD SHARING:
Plan to Share IPD: Undecided